CLINICAL TRIAL: NCT05551663
Title: Isometric Exercise Training in Patients With Heart Failure With Preserved Ejection Fraction: a Randomised Controlled Study
Brief Title: Isometric Exercise Training in Participants With Heart Failure With Preserved Ejection Fraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021.0214
Record Dates: First submitted 2022-09-01; First posted 2022-09-23 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure; Isometric Exercise Training
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric exercise training (Experimental)
  Interventions: Other: Isometric exercise training
- Control group (No Intervention)

INTERVENTIONS:
Other: Isometric exercise training — Participants randomised to the intervention will perform a 4-week programme of isometric exercise training.
  Arms: Isometric exercise training

SUMMARY:
Heart failure with a preserved ejection fraction (HFpEF) is a major cause of morbidity and mortality. Hypertension remains one of the major modifiable risk factors in HFpEF development and progression. The role of aerobic exercise training for blood pressure (BP) reduction is well established, with positive cardiac, vascular, and neurohumoral adaptations all cited as potential mechanisms for improving arterial haemodynamics. However, recent evidence has shown that a specific type of resistance exercise alone, known as isometric exercise (IE), produces greater mean BP reductions than what has traditionally been seen with both aerobic and dynamic resistance exercise training programmes. Indeed, short duration IE training causes significant improvements in both cardiac structure and function, in addition to inducing significant reductions in resting BP in normotensive, pre-hypertensive and hypertensive individuals. This study aims to compare the acute and chronic effects of an IE training intervention on diastolic function parameters in patients who have been diagnosed with HFpEF compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with HFpEF.
* Patients under the care of a St George's Heart Failure cardiology consultant.
* Patients willing and able to provide informed consent.
* Male and female, aged 18 years or above.
* Medically optimised patients.

Exclusion Criteria:

* Recent myocardial infarction or electrocardiographic changes, complete heart block, unstable angina.
* Inability or unwilling to provide informed consent.
* Male and female, aged 17 years or younger.
* Patients with HFrEF.
* Patients with musculoskeletal injury that could conceivably be affected by their involvement.
* Resting BP values of ≥180/110 mmHg.
* Patients unable to understand verbal and written English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Diastolic function | 1-year
  Whether an isometric exercise training (IET) programme statistically significantly improves diastolic function parameters in patients who have been diagnosed with HFpEF. These parameters will be measured quantitatively using transthoracic echocardiography and using measures of transmitral filling velocity (early [E] and late [A] left ventricular filling velocities), the E/A ratio and tissue Doppler velocities (mitral annulus velocities in diastole [E']) and the E/E' ratio.

SECONDARY OUTCOMES:
Blood pressure | 1-year
  Isometric exercise training has been shown to reduce systolic and diastolic blood pressure (mmHg). Our secondary outcome measure is to record any statistically significant changes in blood pressure following a programme of isometric exercise training compared to a control group.

IPD SHARING:
Plan to Share IPD: Undecided